CLINICAL TRIAL: NCT04799847
Title: A Multicenter, Non-randomized, Uncontrolled, Open-label Phase I/II Study to Observe the Safety and Preliminary Efficacy of Catumaxomab in Patients With Non-Muscle-Invasive Bladder Cancer Who Have Failed or Are Intolerant to BCG Vaccine
Brief Title: Catumaxomab in Patients With Non-Muscle-Invasive Bladder Cancer Who Have Failed or Are Intolerant to BCG Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LintonPharm Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LP0190512
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Failed or are Intolerant to BCG Vaccine; catumaxomab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catumaxomab (Experimental): In the dose escalation phase, 2 dose levels of catumaxomab will be explored.
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — This study is conducted in 3 phases sequentially: dose escalation phase, dose expansion phase and dose extension phase. In the dose escalation phase, the preliminary safety and pharmacokinetic profile of catumaxomab by instillation, at 2 dose levels(20ug group and 100ug group）, in NMIBC patients are investigated.

SUMMARY:
A Multicenter, Non-randomized, Uncontrolled, Open-label Phase I/II study to Observe the Safety and Preliminary Efficacy of Catumaxomab in Patients with Non-Muscle-Invasive Bladder Cancer who have Failed or are Intolerant to Bacillus Calmette-Guerin (BCG) Vaccine

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, uncontrolled, open-label phase I/II study to observe the safety and preliminary efficiency of catumaxomab in patients (hereinafter referred to as participants) with non-muscle-invasive bladder cancer (NMIBC) who have failed or are intolerant to Bacillus Calmette-Guerin (BCG) vaccine.

This study is conducted in 3 phases sequentially: dose escalation phase, dose expansion phase and dose extension phase. In the dose escalation phase, the preliminary safety and pharmacokinetic profile of catumaxomab for 4 cycles of instillation in 20ug group participants and 2cycles of instillation in 100ug group participants are explored. Data will be collected after completing DLT observation in all cohorts, but it is not required to lock database. DSMB will review the data of each dose cohort and decide whether to open the enrollment for the next cohort. DSMB will recommend the dose at dose expansion phase according to the relevant data after the completion of DLT observation and the first efficiency assessment.

In the dose expansion phase, 24 participants will receive the catumaxomab treatment at dosing scheme recommended by the DSMB. DLT events occurred within 28 days after the initial instillation will be investigated. After th DLT observation period, DSMB will evaluate the data from both dose escalation and dose expansion phase and decide whether to initiate the dose extension phase; protocol amendment might be developed.

In the dose extension phase, the elgible participants are enrolled and allocated into three arms according to the type of BCG treatment failure: refractory, relapse, and intolerance. A maximum 125 participants are enrolled in the 3 arms, with at least 30 participants allocated to each.

The participants will have chest and abdominal CT and pelvic MRI scan at baseline to determine the area of lesion and to rule out possible extra-bladder lesions. From the initial instillation, cystoscopy, bladder biopsy, urinary cytology, and pelvic MRI scan are performed every 12 weeks (±7 days); chest and abdominal CT scans are performed every 24 weeks (±7 days)1 until recurrence, progression, consent withdrawal, or 96 weeks (±7 days) from the initial instillation, whichever occurs firstly. Participants who discontinue study treatment early due to any reasons other than disease progression will continue to have the tumor response assessment as planned until the participant has disease progression, withdrawal of consent, loss of follow-up, death, 96 weeks (± 7 days) after the initial instillation or until the end of the study, whichever occurs firstly.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent forms have been provided.
2. Willing to be complaint with the study procedures during the study.
3. Male or female, age ≥ 18 years old when signing informed consents.
4. Histologically or cytologically diagnosed as NMIBC, i.e., bladder cancer in the following pTNM status: pTis, pTa, pT1.
5. Have received the standard therapy recommended in the current NMIBC clinical guidelines, including intravesical BCG instillation, and diagnosed as BCG failure or intolerance.
6. Participants had completed TURBT or cystoscopy as required by guidelines prior to enrollment, and no significant tumours were seen in the surgical field Residual lesions
7. Recovered from any toxicity due to previous treatment (Grade 0-1 according to NCI-CTCAE v 5.0).
8. Estimated life span is ≥ 6 months.
9. Eastern Oncology Cooperative Group (ECOG) performance status 0-1.
10. The laboratory test values during the screening period are in accordance with the following table:

    * ANC(absolute neutrophil count)>=1.5x10^9/L
    * Hemoglobin>=80 g/L
    * Platelet>=100x10^9/L
    * Lymphocyte percentage>=20%
    * Serum Bilirubin <=1.25
    * ULN(or 2.5 ULN if there is Gilbert)
    * AST and ALT <=2.5 ULN without liver metastasis（or<=5 ULN if liver metastasis)
    * Serum creatinine <=2.0 mg/dL or
    * Calculated creatinine clearance>=30 mL/min.
11. For women of childbearing potential: use an efficient method for contraception at least 1 month prior to screening and agree to use this method for contraception during the study period and 30 days after the last intravesical instillation.;
12. For men with fertility potential: use condoms or other methods to ensure effective contraception for sexual partners from screening to 30 days after the last intravesical instillation.

Exclusion Criteria:

1. Known or suspected of being allergic to catumaxomab or similar antibodies.
2. Besides the TURBT + immediate postoperative infusion chemotherapy for this NMIBC recurrence, participants received other anti-tumor treatments, including other anti-tumor investigational drugs, chemotherapy, immunotherapy, biological agents, hormone therapy, radiation therapy (excluding local radiation therapy for pain relief), etc., the interval between the last instillation and the first intravesical instillation is ≤ 21 days.
3. Tumor metastases outside the bladder confirmed in imaging examination.
4. With other primary malignant tumors diagnosed before the signing of ICF, excluding squamous cell carcinoma in situ of skin or cervical carcinoma in situ without recurrence within 5 years after resection.
5. The following diseases have not been resolved to CTCAE grade 0-1 in 3 days prior to the first instillation:

   * Uncontrolled acute and chronic infections such as pneumonia, biliary infection, hepatitis B virus infection and hepatitis C virus infection, etc.
   * Dyspnea.
   * Acute /chronic renal injury.
   * Nephrotic syndrome.
   * Bladder perforation.
   * Urinary tract obstruction(except benign prostatic hypertrophy).
6. NYHA Class 3 or 4.
7. Related symptoms and signs of cardiovascular diseases have not been resolved to CTCAE grade 0-1: including myocardial infarction, congestive heart failure, and arrhythmia.
8. Known cerebrovascular accidents have not been resolved to CTCAE grade 0-1.
9. History of autoimmune diseases (eg, inflammatory bowel disease, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autologous hemolytic anemia, rheumatoid arthritis, etc.).
10. Patients with known HIV serology positive, hepatitis C infection and/or hepatitis B (Except the patients with positive HepBsAg or core antibody are responding to anti-HBV treatment, they are allowed to participate in the study.

    Notes: HepBsAg-negative patients at screening, or patients are undergoing treatment with interferon-2a [IFN] or peginterferon-2a [Peg-IFN] and hepatitis B virus [HBV] DNA < 2000 international units [IU], or partients who are receiving nucleoside [acid] analogues at screening and HBV DNA below the lower limit of normal [LLN] are eligible to participate in the study.
11. Pregnancy or breastfeeding during study treatment and follow-up period.
12. Patients with confirmed past history of neurological or psychotic disorders, including epilepsy or dementia.
13. Other serious systemic conditions that may limit the participation in this study (e.g. uncontrolled diabetes, cardiovascular and cerebrovascular disease, severe gastrointestinal disease, and renal disease, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose escalation phase and dose expansion phase only: DLT incidence. | 28 days
  Dose Limited Toxicity
1-year recurrence rate since the initial instillation | 1 year
  1-year recurrence rate since the initial instillation

SECONDARY OUTCOMES:
Recurrence rate at 3 months / 6 months / 2 years. | Up to 2 years
  Recurrence rate at 3 months / 6 months / 2 year
PFS | 2 years
  Relapse-free survival
2-year progression rate to MIBC. | 2 years
  2-year progression rate to MIBC.
The incidence and severity of treatment-emergent adverse events (TEAEs) and Serious adverse event（SAE） | 2 years
  The incidence and severity of treatment-emergent adverse events (TEAEs) and Serious adverse event（SAE） during intravesical instillation with catumaxomab are observed according to the National Cancer Institute Common Terminology Standard for Adverse Events (NCI-CTCAE) v5.0.
ADA | 2 years
  the incidence of anti-drug antibodies (ADA) to catumaxomab by intravesical instillation in serum.
Pharmacokinetic parameters-Cmax | 2 years
  Pharmacokinetic parameters Cmax of bladder perfusion of Catumaxomab in plasma and urine
Pharmacokinetic parameters-Cmin | 2 years
  Pharmacokinetic parameters Cmin of bladder perfusion of Catumaxomab in plasma and urine
Pharmacokinetic parameters-AUC | 2 years
  Pharmacokinetic parameters-AUC of bladder perfusion of Catumaxomab in plasma and urine
Pharmacokinetic parameters-t1/2 | 2 years
  Pharmacokinetic parameters-t1/2 of bladder perfusion of Catumaxomab in plasma and urine

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Third Hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Hospital of Tianjin Medical University, Tianjin